CLINICAL TRIAL: NCT02585492
Title: Episodes of Decreased Oxygen Saturation in Newborns in Skin-to-skin Contact: Role of Maternal Position After Delivery. A Randomized Clinical Study.
Brief Title: Effects of Mother Position in Skin-to-skin Contact Newborn on Oxygen Saturation Levels.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Red Salud Materno Infantil y del Desarrollo (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Neonatologia-2014-02
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Neonatal Disorder
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- head-of-bed elevated 15° (Active Comparator): Mother's head-of-bead elevated 15°. Intervention: Head-of-bed elevated 15° during 2 hours after the delivery.
  Interventions: Other: Head-of-bed elevated 15°
- head-of-bed elevated 45° (Experimental): Mother's head-of-bead elevated 45°. Intervention: Head-of-bed elevated 45°during 2 hours after delivery.
  Interventions: Other: Head-of-bed elevated 45°

INTERVENTIONS:
Other: Head-of-bed elevated 15° — Head-of-bed elevated 15° during 2 hours after delivery.
  Arms: head-of-bed elevated 15°
Other: Head-of-bed elevated 45° — Head-of-bed elevated 45° during 2 hours after delivery.
  Arms: head-of-bed elevated 45°

SUMMARY:
The purpose of this study is to determine if the position of the mother in the first two hours after delivery, while she is in skin to skin contact with your child, influences the oxygen saturation and/or heart rate of the newborn. In this way it could provide some useful information for the prevention of seemingly lethal episodes or sudden death of the child when, following current recommendations is skin to skin contact in the first hours of life. These episodes are communicating in all developed countries and have caused great concern and interest in the scientific community. So far we only have information from case series.

DETAILED DESCRIPTION:
The early skin to skin contact between mother and child in the first two hours postpartum is essential for bonding and breastfeeding. Coinciding with the widespread application of this procedure in hospitals have been described, in different countries, cases of children who have suffered episodes of apparent life threatening events (ALTEs) or early sudden deaths during the same procedure. The cause of these events is unclarified, it is unknown whether the position of the mother during the first two hours of a child's life affects their stability.

The investigators's hypothesis is that the frequency of episodes of oxygen saturation less than 91% in the first 2 hours of life of the newborn is reduced by one third in children whose mothers are incorporated at 45° above the horizontal plane of the bed compared with children whose mothers are incorporated to 15º.

This is a multicenter, randomized and controlled study in 10 Spanish hospitals with blind evaluation. 5866 participants will be enrolled in this study (a total of 1275 children are required in each arm of the study).

Mother/child (defined as a dyad) will be randomized in two groups:

Group A: head-of-bed elevated 15°. Group B: head-of-bed elevated 45°.

ELIGIBILITY:
Inclusion criteria:

1. Single fetus pregnancy
2. Pregnancy controlled or partially controlled(1)
3. Normal pregnancy or with gestational diabetes treated with diet, high blood pressure controlled with only a drug as maximum (without preeclampsia)
4. Gestation to term (between 37 weeks to 41 weeks and 6 days of gestational age).
5. Maternal temperature at onset of labor ≤38 degrees Celsius
6. Presence of a companion during the 2 hours after delivery
7. Desire of the mother to perform early skin-to-skin

Exclusion criteria pre-randomization:

1. Consumption of tobacco, alcohol, drugs or any medication with sedative or relaxing(2) effect or any pathology during pregnancy.
2. Prenatal diagnosis of chromosomal abnormalities or major malformations.
3. Prenatal diagnosis of intrauterine growth restriction with any degree of alteration in the flow as well as the abnormal small-for-gestational-age fetuses (due to malformations, intrauterine infection ...).
4. No companion during the first two hours postpartum

Notes:

1. Partially controlled pregnancy: she has the 20 weeks ultrasound but lack the first and/or third trimester of pregnancy and/or analytical (serology, O'Sullivan test ...).
2. Medicinal products with sedative or relaxing effect: opioids, anticonvulsants, antipsychotics, benzodiazepines, anxiolytics, hypnotics, antidepressants and sedative plants.

Post randomization exclusion criteria (at the end of delivery)

1. Related to childbirth:

   * Caesarean section or instrumental delivery (forceps, vacuum)
   * Maternal fever >38 degrees Celsius
   * Mother hemodynamic instability (hypotension, tachycardia, altered level of consciousness, poor perfusion, striking pallor)
   * Cord prolapse
   * Signs of fetal distress with lower pH fetal scalp <7.25 or umbilical artery pH <7.20
   * Any other obstetrical complication
2. Related mother:

   * Any type of illness
   * Sedatives or relaxants during or after birth(3)
3. Related Newborn (RN)

   * Need for resuscitation measures
   * Major malformation diagnosed intrapartum
   * Apgar ≤7 at one minute, 5 or 10 minutes
   * Presence of clinic(4) before the 10 minutes of life
   * Birth weight <2300 g or>4500 g
4. Interruption of skin contact because the mother present a problem

Notes:

(3) Sedatives or relaxants during or after birth: Pethidine (Dolantina®), scopolamine (Buscapina®), haloperidol, benzodiazepines and opiates.

(4) Clinic: general discomfort, fever, hypothermia, pallor, mottled skin (cutis marmorata), cyanosis, petechiae, purpura, lethargy, weakness, poor responsiveness, seizures, tremors, poor perfusion, maintained tachycardia, bradycardia, hypotension, apnea, tachypnea, respiratory distress (grunting, nasal flaring, intercostal or subcostal or substernal retractions, thoracoabdominal dissociation), vomiting, abdominal distesion, etc.

Clarifications:

It can include:

1. Newborns with intrauterine diagnosis of ectasia pyelocaliceal grades I and/or II, choroid plexus cysts, aberrant right subclavian artery or single umbilical artery (minor malformations).
2. Newborns whose time broken bag is ≥ to 18 hours provided that they do not present clinic(4).
3. Newborn with risk of infection without symptoms at birth.
4. Newborn with stained amniotic fluid, born crying, who does not require tracheal aspiration, or resuscitation and shows no clinical(4) signs during the first 10 minutes after birth.
5. Small for normal fetal gestational age (genetic-family origin)

Ages: 259 Days to 293 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1243 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Presence of at least one episode desaturation ≤90% | Two first hours after delivery
  The evaluation will be done with a pulse oximeter (non-invasive Radical-7 Signal Extraction PulseCO-Oximeter equipped with Masimo Rainbow SET technology). All the technology used in all hospitals is part of Masimo's SafeyNet system.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia R. García Lara, Dra, Study Chair — Hospital Universitario 12 de Octubre
Locations (7):
- Spain (7):
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de Cruces, Bilbao, Vizcaya
  - Hospital de Vielha, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Quirón, Madrid
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez Lopez J, Garcia Lara NR, Lopez Maestro M, De la Cruz Bertolo J, Martinez Avila JC, Vento M, Parra Llorca A, Izquierdo Macian I, Pellicer A, Marin Huarte N, Asla Elorriaga I, Roman Echevarria L, Copons Fernandez C, Martin Ancel A, Cabanas F, Garcia Algar O, Pallas Alonso CR. What is the impact of mother's bed incline on episodes of decreased oxygen saturation in healthy newborns in skin-to-skin contact after delivery: Study protocol for a randomized controlled trial. Trials. 2019 Mar 20;20(1):179. doi: 10.1186/s13063-019-3256-0. PMID 30894206